CLINICAL TRIAL: NCT00152477
Title: A Two-Part, Open Label Phase II Trial: Part One, Dose Escalation Safety; Part Two, Randomized/Comparing CDP791 Plus Carboplatin/Paclitaxel With Carboplatin/Paclitaxel Alone in Subjects With Locally Advanced or Metastatic Non-Squamous Non-Small-Cell Lung Cancer
Brief Title: A Study of Paclitaxel/Carboplatin With or Without CDP791 in Patients With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C79102
Record Dates: First submitted 2005-09-06; First posted 2005-09-09 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma; Non-Squamous Non-Small-Cell Lung Cancer
Keywords: Non-small-cell-lung cancer; carboplatin; paclitaxel; VEGF; monoclonal antibody
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

ARMS (3):
- Carboplatin/Paclitaxel (Experimental): Carboplatin and paclitaxel alone.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Carboplatin/Paclitaxel/CDP791 10mg (Experimental): Carboplatin and paclitaxel plus CDP791 10mg/kg
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: CDP791 10mg/kg; Drug: CDP791 20mg/kg
- Carboplatin/Paclitaxel/CDP791 20mg (Experimental): Carboplatin and paclitaxel plus CDP791 20mg/kg
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: CDP791 10mg/kg; Drug: CDP791 20mg/kg

INTERVENTIONS:
Drug: Carboplatin — 10mg/mL vial AUC6. Dosed intravenously over 15-30 minutes immediately following paclitaxel, Day 0 of each cycle.
  Each cycle to be repeated every three weeks for a maximum of six cycles.
  Other Names: CBDCA, Paraplatin, JM-8, NSC 241240
Drug: Paclitaxel — 6mg/mL vial 200 mg/m2 iv over three hours, Day 0. Each cycle to be repeated every 3 weeks for a maximum of 6 cycles.
  Other Names: Taxol, NSC #673089
Drug: CDP791 10mg/kg — CDP791 20mg/mL vial CDP791 diluted (10mg/kg or 20mg/kg) in 0.9% saline will be given as a 200mL iv infusion over approximately 60 minutes following administration of standard chemotherapy.
  Arms: Carboplatin/Paclitaxel/CDP791 10mg; Carboplatin/Paclitaxel/CDP791 20mg
Drug: CDP791 20mg/kg — CDP791 20mg/kg CDP791 diluted (10mg/kg or 20mg/kg) in 0.9% saline will be given as a 200mL iv infusion over approximately 60 minutes following administration of standard chemotherapy.
  Arms: Carboplatin/Paclitaxel/CDP791 10mg; Carboplatin/Paclitaxel/CDP791 20mg

SUMMARY:
A 2-part study to examine safety, tolerability and pharmacokinetics (part 1), and anti-tumour effects (part 2), of CDP791 combined with carboplatin and paclitaxel.

DETAILED DESCRIPTION:
This is a two part study to investigate the safety and anti-tumour effects of standard chemotherapy, plus an investigational drug (CDP791), in patients with advanced non small cell lung cancer.

In part one, patients receive carboplatin and paclitaxel chemotherapy together with one of 2 doses of CDP791. The main aim of this part is to investigate safety and tolerability of carboplatin/paclitaxel plus CDP791.

If part one confirms that the combination of drugs is safe and well tolerated, 156 patients will enter part 2. They will be randomized to receive either carboplatin/paclitaxel (C/P) alone, or C/P plus one of 2 doses of CDP791. The main aim of this part of the study is to compare the anti-tumor effects of CDP791 plus C/T with those of C/T alone. Participants will receive up to six cycles of chemotherapy with or without CDP791. Those whose disease stabilizes, or responds, will be eligible to continue to receive CDP791. Participants in the C/T alone arm whose disease progresses will be eligible to receive CDP791 monotherapy.

Participants will be followed up longterm, so that survival can be measured.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Male and female subjects with Stage IIIb (with malignant pleural effusion or if no pleural effusion is present subjects who are not candidates for combined modality therapy), Stage IV, or recurrent non-squamous, non-small-cell lung carcinoma.
* The subject must be aged 18 years or above.
* The subject must have ECOG performance status of 0 or 1 and a life expectancy of at least three months.
* Subjects will have measurable disease.
* The subject must be able to understand the information provided to them and to give written informed consent.
* Female subjects must be either postmenopausal, surgically sterilized, or using a method of contraception judged reliable by the Investigator.
* Male subjects must be using a method of contraception judged reliable by the Investigator.

Exclusion Criteria:

* Subjects with squamous cell lung carcinoma.
* Subjects with lung lesions located centrally in the chest that involve major blood vessels.
* Concurrent active malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix. Subjects with previous malignancies are eligible provided that they have been disease free for five years or more.
* Presence of additional major chronic disease such as hepatic or renal dysfunction, cardiac dysfunction, peripheral vascular disease, evidence of a myocardial infarction within six months of Screening visit, tuberculosis or epilepsy.
* Subjects known to be infected with hepatitis B or C virus or HIV 1 or 2.
* Any evidence of serious active infection (ie requiring an iv antibiotic or antiviral agent).

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-08-15 (Actual); Primary Completion 2009-06-25 (Actual); Study Completion 2009-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (21):
- Hungary (5):
  - Budapest
  - Deszk
  - Mátraháza
  - Nyíregyháza
  - Pécs
- Poland (12):
  - Krakow
  - Lodz
  - Lublin
  - Olsztyn
  - Otwock
  - Poznan
  - Radom
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
  - Zabrze
- Russia (4):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Samara

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in August 2005 and concluded in June 2009. Across Part I (dose escalation) and Part II (Open Label randomized) of the study, 165 subjects were analyzed. Part II was opened for 156 response-evaluable subjects.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Period: Chemotherapy Period
Arm/Group | Carboplatin/Paclitaxel | Carboplatin/Paclitaxel/CDP791 10mg | Carboplatin/Paclitaxel/CDP791 20mg
Started | 50 | 56 | 59
Part II | 50 | 53 | 53
Completed | 22 | 34 | 39
Not Completed | 28 | 22 | 20
Not completed — Adverse Event | 9 | 4 | 5
Not completed — Death | 1 | 3 | 3
Not completed — Lack of Efficacy | 4 | 5 | 6
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Progression of Disease | 6 | 8 | 4
Not completed — Investigator decision | 0 | 0 | 1
Not completed — Patient condition worsened | 1 | 0 | 0
Period: Monotherapy Period
Arm/Group | Carboplatin/Paclitaxel | Carboplatin/Paclitaxel/CDP791 10mg | Carboplatin/Paclitaxel/CDP791 20mg
Started | 15 (7 subjects completed the Chemotherapy period but did not enter the Monotherapy period.) | 29 (5 subjects completed the Chemotherapy period but did not enter the Monotherapy period.) | 34 (5 subjects completed the Chemotherapy period but did not enter the Monotherapy period.)
Part II | 13 | 26 | 29
Completed | 0 | 0 | 0
Not Completed | 15 | 29 | 34
Not completed — Adverse Event | 1 | 0 | 5
Not completed — Death | 2 | 0 | 1
Not completed — Lack of Efficacy | 7 | 16 | 10
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Progression of Disease | 5 | 11 | 12
Not completed — Patient decision | 0 | 1 | 1
Not completed — Study personel decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to all response-evaluable Part II subjects.
Arm/Group | Carboplatin/Paclitaxel | Carboplatin/Paclitaxel/CDP791 10mg | Carboplatin/Paclitaxel/CDP791 20mg | Total Title
Number analyzed (Participants) | 50 | 53 | 53 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 35 | 40 | 105
  >=65 years | 20 | 18 | 13 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.58 (10.69) | 60.70 (10.01) | 58.25 (9.38) | 60.15 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 29 | 70
  Male | 30 | 32 | 24 | 86

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (RR)
Description: Participants are evaluated for response using Response Evaluation Criteria in Solid Tumors (RECIST) (Therasse P et al; 2000). The tumor response rate is calculated as the total number of subjects whose best overall response is a complete response (CR)= disappearance of all target lesions; or a partial response (PR) = >=30 % decrease in the sum of the longest diameter of target lesions, divided by the number of randomized subjects (RS):
  (CR + PR) / RS.
Time Frame: 24 weeks
Population: All Randomized Part II Subjects
Measure: Number; unit: percentage of participants
Groups:
- Carboplatin/Paclitaxel (Randomized Part II SjS): Carboplatin and paclitaxel alone (Randomized Part II Subjects Set [SjS])
- Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS): Pooled CDP791 10 mg/kg or 20 mg/kg + CT treatment arms
- Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS): Carboplatin and paclitaxel plus CDP791 10mg/kg (Randomized Part II Subjects Set [SjS])
- Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS): Carboplatin and paclitaxel plus CDP791 20mg/kg (Randomized Part II Subjects Set [SjS])
Arm/Group | Carboplatin/Paclitaxel (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS) | Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS)
Number analyzed (Participants) | 50 | 106 | 53 | 53
percentage of participants
  Complete responder | 0 | 0 | 0 | 0
  Partial responder | 20 | 26.4 | 22.6 | 30.2
Statistical Analysis 1: Comparison: Carboplatin/Paclitaxel (Randomized Part II SjS) vs Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS); Test type: Superiority; p = 0.384, Cochran-Mantel-Haenszel — Two-sided Chi-square test. Fisher's Exact test presented when number of responders in a treatment group is <5; Difference of response rate = 6.4, 95% CI 2-sided [-7.7 to 20.5]
Statistical Analysis 2: Comparison: Carboplatin/Paclitaxel (Randomized Part II SjS) vs Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS); Test type: Superiority; p = 0.409, Cochran-Mantel-Haenszel — CMH test stratified by country and disease stage (3 levels: Stage IIIb without malignant pleural effusion versus Stage IIIb with malignant pleural effusion or Stage IV or recurrent); Difference of response rate = 6.4, 95% CI [-7.7 to 20.5]
Statistical Analysis 3: Comparison: Carboplatin/Paclitaxel (Randomized Part II SjS) vs Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS); Test type: Superiority; p = 0.744, Chi-squared — Two-sided Chi-square test. Fisher's Exact test presented when number of responders in a treatment group is < 5; Difference of response rate = 2.6, 95% CI 2-sided [-13.5 to 18.8]
Statistical Analysis 4: Comparison: Carboplatin/Paclitaxel (Randomized Part II SjS) vs Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS); Test type: Superiority; p = 0.783, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Difference of response rate = 2.6, 95% CI 2-sided [-13.5 to 18.8]
Statistical Analysis 5: Comparison: Carboplatin/Paclitaxel (Randomized Part II SjS) vs Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS); Test type: Superiority; p = 0.234, Chi-squared — Two-sided Chi-square test. Fisher's Exact test presented when number of responders in a treatment group is < 5; Difference of response rate = 10.2, 95% CI 2-sided [-6.8 to 27.2]
Statistical Analysis 6: Comparison: Carboplatin/Paclitaxel (Randomized Part II SjS) vs Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS); Test type: Superiority; p = 0.228, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Difference of response rate = 10.2, 95% CI 2-sided [-6.8 to 27.2]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as time from date of randomization until the date progressive disease (PD) is first recorded or until death, whichever is first.
Time Frame: Up to 57 weeks
Population: All Randomized Part II Subjects
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS): Carboplatin and paclitaxel plus CDP791 10mg/kg (Randomized Part II Subjects Set [SS])
Arm/Group | Carboplatin/Paclitaxel (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS) | Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS)
Number analyzed (Participants) | 50 | 106 | 53 | 53
weeks | 24.14 [20.29 to 29.29] | 26.86 [24.43 to 30.14] | 26.86 [21.14 to 30.71] | 25.43 [24.29 to 30.43]

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) is defined as the time from date of randomization until the date of progression, death or, for subjects who discontinued treatment for toxicity reason, their last dosing date, whichever occurs first.
Time Frame: Up to 57 weeks
Population: All Randomized Part II Subjects
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Carboplatin/Paclitaxel (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS) | Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS)
Number analyzed (Participants) | 50 | 106 | 53 | 53
weeks | 13.21 [6.86 to 20.29] | 21.71 [18.14 to 24.71] | 18.43 [12.14 to 24.71] | 24.29 [18.14 to 27.00]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of randomization until the date of death.
Time Frame: Up to 57 weeks
Population: All Randomized Part II Subjects
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Carboplatin/Paclitaxel (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS) | Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS)
Number analyzed (Participants) | 50 | 106 | 53 | 53
weeks | 36.14 [27.14 to 64.14] | 47.14 [40.43 to 56.00] | 46.57 [38.57 to 59.86] | 47.57 [31.29 to 75.00]

5. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response is measured from the time measurement criteria are first met for complete response (CR) or partial response (PR), whichever is recorded first, until the first date of documented progressive disease or death.
Time Frame: Up to 57 weeks
Population: The duration of overall response was computed for subjects only, whose best response was either PR or CR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Carboplatin/Paclitaxel (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS) | Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS)
Number analyzed (Participants) | 10 | 28 | 12 | 16
weeks | 21.14 [19.14 to NA] — Upper limit is not estimable due to insufficient number of responding patients who later go on to disease progression or death. | 21.14 [16.86 to 22.43] | 21.14 [19.29 to NA] — Upper limit is not estimable due to insufficient number of responding patients who later go on to disease progression or death. | 18.00 [16.71 to 22.43]

6. Secondary Outcome: Time to Response
Description: Time to response is defined as the time from the first dose of study therapy until measurement criteria are first met for complete response or partial response (whichever is recorded first).
Time Frame: Week 24
Population: The time to response was computed for subjects only, whose best response was either PR or CR.
Measure: Median (Full Range); unit: weeks
Arm/Group | Carboplatin/Paclitaxel (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 (Randomized Part II SjS) | Carboplatin/Paclitaxel/CDP791 10mg (Randomized Part II SS) | Carboplatin/Paclitaxel/CDP791 20mg (Randomized Part II SjS)
Number analyzed (Participants) | 10 | 28 | 12 | 16
weeks | 8.57 [8.14 to 17.43] | 9.14 [8.36 to 16.64] | 11.86 [8.86 to 16.64] | 9.00 [8.21 to 15.29]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 1 until Safety Follow-Up Visit (for up to 57 weeks).
Description: All Treated Subjects: all subjects who took at least one dose of study drug.
Groups:
- Carboplatin/Paclitaxel (SS): Carboplatin and paclitaxel alone.
- Carboplatin/Paclitaxel/CDP791 (SS): Pooled CDP791 10 mg/kg or 20 mg/kg + CT treatment arms
- Carboplatin/Paclitaxel/CDP791 10mg (SS): Carboplatin and paclitaxel plus CDP791 10mg/kg
- Carboplatin/Paclitaxel/CDP791 20mg (SS): Carboplatin and paclitaxel plus CDP791 20mg/kg
Arm/Group | Carboplatin/Paclitaxel (SS) | Carboplatin/Paclitaxel/CDP791 (SS) | Carboplatin/Paclitaxel/CDP791 10mg (SS) | Carboplatin/Paclitaxel/CDP791 20mg (SS)
All-Cause Mortality (participants affected / at risk) | 30/50 | 72/115 | 39/56 | 33/59
Serious Adverse Events (participants affected / at risk) | 18/50 | 36/115 | 18/56 | 18/59
Other Adverse Events (participants affected / at risk) | 44/50 | 110/115 | 54/56 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Paclitaxel (SS) (N=50) | Carboplatin/Paclitaxel/CDP791 (SS) (N=115) | Carboplatin/Paclitaxel/CDP791 10mg (SS) (N=56) | Carboplatin/Paclitaxel/CDP791 20mg (SS) (N=59)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 2 | 4
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5 | 2 | 3
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0
Condition aggravated (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 2
General physical health deterioration (General disorders) | 0 | 2 | 1 | 1
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Injection site abscess (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Scan abnormal (Investigations) | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 1 | 3 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 1
Metastases to mouth (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 3
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Paclitaxel (SS) (N=50) | Carboplatin/Paclitaxel/CDP791 (SS) (N=115) | Carboplatin/Paclitaxel/CDP791 10mg (SS) (N=56) | Carboplatin/Paclitaxel/CDP791 20mg (SS) (N=56)
Anaemia (Blood and lymphatic system disorders) | 17 | 35 | 17 | 18
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 5 | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 23 | 14 | 9
Neutropenia (Blood and lymphatic system disorders) | 15 | 42 | 19 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 19 | 8 | 11
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 4 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 9 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 7 | 16 | 6 | 10
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 3 | 1
Vomiting (Gastrointestinal disorders) | 8 | 9 | 5 | 4
Asthenia (General disorders) | 3 | 9 | 4 | 5
Chest pain (General disorders) | 4 | 9 | 5 | 4
Fatigue (General disorders) | 10 | 16 | 9 | 7
Oedema peripheral (General disorders) | 3 | 10 | 5 | 5
Pyrexia (General disorders) | 2 | 8 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 6 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 2 | 5 | 2 | 3
Blood creatinine increased (Investigations) | 1 | 5 | 2 | 3
Blood glucose increased (Investigations) | 2 | 12 | 8 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 8 | 4 | 4
Weight decreased (Investigations) | 3 | 6 | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 6 | 18 | 8 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 14 | 4 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 15 | 6 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 0
Neuropathy (Nervous system disorders) | 3 | 4 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 4 | 1 | 3
Paraesthesia (Nervous system disorders) | 5 | 5 | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 12 | 7 | 5
Polyneuropathy (Nervous system disorders) | 2 | 4 | 1 | 3
Insomnia (Psychiatric disorders) | 3 | 4 | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 9 | 3 | 6
Proteinuria (Renal and urinary disorders) | 1 | 13 | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 4 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 38 | 19 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0
Hypertension (Vascular disorders) | 1 | 12 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days